CLINICAL TRIAL: NCT04529850
Title: An Open Label Multi-Center Study of the Effects of GC4419 When Administered to Reduce the Incidence and Severity of Severe Oral Mucositis Associated With Chemo RT for Locally Advanced, Non-Metastatic Head and Neck Cancer
Brief Title: Ph 2 Open Label Study of GC4419 to Reduce SOM Associated With Chemoradiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GTI-4419-202
Record Dates: First submitted 2020-08-13; First posted 2020-08-28 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer; Oral Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — avasopasem manganese; Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Intervention Model Description: To evaluate the effects of GC4419 in subjects with head and neck cancer, who are at high risk for Severe Oral Mucositis (SOM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Active Arm (Experimental): 90mg GC4419 by IV
  Interventions: Drug: Drug: GC4419; Radiation: Intensity-modulated radiation therapy (IMRT); Drug: Cisplatin

INTERVENTIONS:
Drug: Drug: GC4419 — GC4419 60 Minute Infusion
Radiation: Intensity-modulated radiation therapy (IMRT) — 2.0 to 2.2 Gy daily over 7 weeks
Drug: Cisplatin — 100mg/m2 once every 3 weeks or 40mg/m2 once weekly for 6-7 doses

SUMMARY:
GTI-4419-202 is a Phase 2 open-label study of the effects of GC4419 (IV) when administered in combination with IMRT and cisplatin to up to subjects with head and neck cancer, who are at high risk for Severe Oral Mucositis (SOM)

DETAILED DESCRIPTION:
Subjects will receive 90 mg GC4419 per day (60 min IV infusion to complete within 60 minutes prior to IMRT), concurrent with daily fractions of IMRT (2.0-2.2 Gy) to a total of 60-72 Gy over approximately 7 weeks, plus cisplatin administered 100 mg/m2 once every three weeks for 3 doses or 40 mg/m2 once weekly for 6-7 doses (Investigator's choice).

All subjects will be assessed twice weekly for Oral Mucositis (OM) per WHO grading criteria until 28 days post end of study treatment period (last day of IMRT).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically-confirmed diagnosis of locally advanced squamous cell carcinoma of the head and neck that will be treated with cisplatin plus concurrent IMRT.
2. Treatment plan to receive a continuous course of IMRT delivered as single daily fractions of 2.0 to 2.2 Gy with a cumulative radiation dose of 60-72 Gy.
3. Patients who have had prior surgery may be eligible,
4. Treatment plan to receive standard cisplatin monotherapy administered either every three weeks (100 mg/m2 for 3 doses) or weekly (40 mg/m2 for 6-7 doses).
5. Age 18 years or older
6. ECOG performance status ≤ 2
7. Adequate hematologic function
8. Adequate renal and liver function Alkaline phosphatase ≤ 2.5 ULN

Exclusion Criteria:

1. Metastatic disease
2. Prior radiotherapy to the region of the study cancer or adjacent anatomical sites
3. Prior induction chemotherapy or plans for chemotherapy to be administered only sequentially with IMRT
4. Planned concurrent chemotherapy other than single agent cisplatin
5. Receiving any approved or investigational anti-cancer agent
6. Concurrent participation in another interventional clinical study
7. Inability to eat soft solid food at baseline for reasons other than mouth soreness after surgery or dental procedures
8. Complete reliance on parenteral or gastrointestinal tube-delivered nutrition at baseline
9. Malignant tumors other than head and neck cancer (HNC) within the last 5 years
10. Active infectious disease excluding oral candidiasis
11. Presence of oral mucositis at baseline.
12. Known history of human immunodeficiency virus (HIV) or active hepatitis B/C
13. Female patients who are pregnant or breastfeeding
14. Known allergies or intolerance to cisplatin and similar platinum-containing compounds
15. Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating Investigator, create a risk for a precipitous decrease in blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Holmlund, MD, Study Chair — Chief Medical Officer
Locations (24):
- Belgium (4):
  - Onze-Lieve-Vrouwziekenhuis (OLVZ) - Campus Aalst, Aalst
  - AZ Klina, Brasschaat
  - Az Nikolaas, Sint-Niklaas
  - CHR Verviers, Verviers
- Fakultni Nemocnice Na Bulovce, Prague, Czechia
- Germany (2):
  - University Medical Center Schleswig-Holstein, Kiel
  - Universitatsklinikum Leipzig AoR, Leipzig
- Poland (4):
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - Szpitale Pomorskie Sp. z o.o., Pomorskie
  - Cancer Center Institute of Oncology, Warsaw
- Spain (11):
  - Complejo Hospitalario Universitario De Santiago De Compostela, A Coruña
  - Gurutzetako Unibersitate Ospitalea - Hospital Universitario Cruces - Instituto BioCruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Institut Catala d'Oncologia de Girona, Girona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Madrid Universitario Sanchinarro (Centro Integral Oncologico Clara Campal), Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Complejo Hospitalario de Navarra (CHN), Pamplona
  - Hospital universitario Virgen del Rocio, Salamanca
  - Universidad de Salamanca - Hospital Clinico Universitario, Salamanca
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital of Bern, Inselspital, Fribourg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 subjects were enrolled to the study (signed an ICF). Only 37 of these subjects were dosed on the trial and part of the ITT population (enrolled subjects who received 1 dose of study medication). The 1 subject that was enrolled but was not dosed withdrew their consent prior to treatment.
Period: Overall Study
Arm/Group | Open Label Active Arm
Started | 37
Completed | 32
Not Completed | 5
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Active Arm
Number analyzed (Participants) | 37
Age, Customized [Count of Participants; unit: Participants]
  Age Group, years: <18 | 0
  Age Group, years: 18-65 | 25
  Age Group, years: 66-75 | 10
  Age Group, years: >75 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 8
  Czechia | 4
  Poland | 8
  Switzerland | 7
  Germany | 1
  Spain | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent AE's
Description: Number of Subjects with at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: First dose of study medication through the 30 days following the last dose of IMRT, GC4419, or cisplatin (whichever occurs last) which is estimated to be 11 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Active Arm
Number analyzed (Participants) | 37
Participants
  TEAE | 36
  TEAE Related to GC4419 | 12
  TEAE Related to IMRT | 33
  TEAE Related to Chemotherapy | 35
  TEAE Leading to Discontinuation | 11
  TEAE Leading to Discontinuation of GC4419 | 1
  TEAE Leading to Discontinuation of IMRT | 1
  TEAE Leading to Discontinuation of Chemotherapy | 10

2. Secondary Outcome: Cumulative Incidence of Severe OM
Description: Cumulative Incidence of WHO Grade 3-4 from the start of IMRT through the end of the study treatment period (last day of IMRT)
Time Frame: From start of Intensity-modulated radiation therapy (IMRT) through approximately 30 fractions which is estimated to be 6-7 weeks.
Population: Per Protocol Population defined as subjects who received at least 60 Gy of IMRT and at least 25 doses of GC4419.
Measure: Number (95% Confidence Interval); unit: percentage of Subjects with SOM
Arm/Group | Open Label Active Arm
Number analyzed (Participants) | 33
percentage of Subjects with SOM | 54.5 [36.35 to 71.89]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the first administration of study drug through 30 days following the last dose of IMRT, cisplatin, or study drug (whichever occurred last) which is estimated to be 11 weeks
Arm/Group | Open Label Active Arm
All-Cause Mortality (participants affected / at risk) | 2/37
Serious Adverse Events (participants affected / at risk) | 18/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Active Arm (N=37)
Pneumonia (Infections and infestations) | 3 (3)
COVID 19 (Infections and infestations) | 2 (2)
Device Related Infection (Infections and infestations) | 1 (1)
Stoma Site Infection (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leuokopenia (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Tumor Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Active Arm (N=37)
Nausea (Gastrointestinal disorders) | 19 (23)
Constipation (Gastrointestinal disorders) | 10 (12)
Dysphagia (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 8 (11)
Diarrhoea (Gastrointestinal disorders) | 7 (11)
Dyspepsia (Gastrointestinal disorders) | 6 (12)
Dry Mouth (Gastrointestinal disorders) | 5 (7)
Oral Pain (Gastrointestinal disorders) | 5 (8)
Lymphopenia (Blood and lymphatic system disorders) | 25 (32)
Leukopenia (Blood and lymphatic system disorders) | 15 (20)
Anaemia (Blood and lymphatic system disorders) | 14 (19)
Neutropenia (Blood and lymphatic system disorders) | 10 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (9)
Hypomagnesamia (Metabolism and nutrition disorders) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9)
Asthenia (General disorders) | 7 (13)
Pyrexia (General disorders) | 7 (11)
Oral Candidiasis (Infections and infestations) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 7 (9)
Weight Decreased (Investigations) | 5 (6)
Hypotension (Vascular disorders) | 7 (8)
Radiation Skin Injury (Injury, poisoning and procedural complications) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI has publication and presentation privileges provided that manuscript/presentation is submitted to the sponsor 60 days prior to submission of the publication or 60 days prior to presentation. PI agrees to remove confidential information of sponsor prior to submission of publication or presentation or defer submission until confidential information can be protected by filing of a patent application. PI cannot publish the results from their site until the sponsor has published multi-site data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04529850/Prot_SAP_000.pdf